CLINICAL TRIAL: NCT05840874
Title: Surgical Complications of Enterocystoplasty in Children: A Retrospective Monocentric Study About 39 Cases
Brief Title: Complications of Enterocystoplasty in Children
Acronym: AVPED
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dr Christelle DESTINVAL (Other)
Responsible Party: Sponsor-Investigator, Dr Christelle DESTINVAL, Principal Investigator, University of Lorraine
Organization: University of Lorraine (Other)
Other Study IDs: ULorraine; 2021PI090 (Registry Identifier: DRCI)
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Complications of Surgical Procedure; Neurogenic Bladder; Spina Bifida; Child, Only
Keywords: Augmentation Enterocystoplasty; Surgical Complications; Children; Retrospective Study
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Dysraphism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to describe the complications in participants who underwent enterocystoplasty in childhood.

The main question[s] it aims to answer are:

* what kind of complications are there
* the kind of complications depending on the type of enterocystoplasty Participants data will be collected in the medical field. There is no comparison group.

DETAILED DESCRIPTION:
From 1982 to 2020, all patients who had an enterocystoplasty in childhood were collected.

Complications were numbered depending on the type of enterocystoplasty and the investigators tried to find which risk factors exist.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent a enterocystoplasty before 18 years old

Exclusion Criteria:

* patients who underwent a enterocystoplasty after 18 years old

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with dysfunctional bladder
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Surgical complications of bladder augmentation in children depending on the type of enterocystoplasty | 38 years
  Observational study

SECONDARY OUTCOMES:
Impact of the participants' age on the occurrence of complications depending on the type of enterocystoplasty | 38 years
  Observational study
Impact of the participants' sex on the occurrence of complications depending on the type of enterocystoplasty | 38 years
  Observational study
Impact of the participants' type of neurogenic bladder on the occurrence of complications depending on the type of enterocystoplasty | 38 years
  Observational study: the participants can have spina bifida, bladder exstrophy, anorectal malformation and if it has an impact on the occurrence of complications depending on the type of enterocystoplasty

CONTACTS AND LOCATIONS:
Locations (1):
- ULorraine, Nancy, France

IPD SHARING:
Plan to Share IPD: No
In the name of anonymization we won't share individual participant data

REFERENCES:
- [Background] Molina CA, Lima GJ, Cassini MF, Andrade MF, Facincani I, Tucci Junior S. Complications after bladder augmentation in children. Acta Cir Bras. 2016;31 Suppl 1:8-12. doi: 10.1590/S0102-86502016001300003. PMID 27142898